CLINICAL TRIAL: NCT03157518
Title: Oral Probiotic Administration to Modulate the Airway Microbiome in Obese Asthmatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jennifer Trevor, Assistant Professor of Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F170105003
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Asthma; obesity; micorbiome; probiotics
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients enrolled will receive probiotic supplementation following the first bronchoscopy for four weeks. A second bronchoscopy will be performed following probiotic administration.
  Interventions: Dietary Supplement: Seeking Health Probiota Bifido

INTERVENTIONS:
Dietary Supplement: Seeking Health Probiota Bifido — • This is a proof of concept study to demonstrate that oral probiotic use can modulate the airway microbiome. After informed consent has been obtained, this study will consist of 2 visits over a four week time period. Each visit will include a blood draw (30ml) and a research bronchoscopy/ bronchoalveolar lavage (BAL) (200ml) visit . A urine pregnancy test will be done on all females of childbearing potential prior to the first BAL as well as a CBC, BMP, and blood clotting tests in all participants. Following the first BAL, subjects will be asked to take an over the counter probiotic supplement (Seeking Health Probiota Bifido) nightly which will be provided to the participant by the study coordinator until the 2nd BAL is performed 4 weeks after the first BAL.

SUMMARY:
Obesity is a major health concern in the Deep South resulting in a growing number of metabolic disorders that strain the resources of our healthcare system. Obesity is recognized as a major risk factor for asthma. The Centers for Disease Control and Prevention (CDC) has stated "obesity is associated significantly with the development of asthma, worsening asthma symptoms, and poor asthma control. This leads to increased medication use and hospitalizations."

Variations in the airway microbiome are correlated with the risk for development of asthma, and populations of different bacteria vary by phenotype amongst severe asthmatics . Proteobacteria are found in greater proportion in asthmatic subjects relative to healthy controls (37% vs 15%) while non-asthmatic subjects have a relative abundance of Firmicutes (47% vs 63%) and Actinobacteria (10% vs 14%) compared to those with asthma . Amongst those with asthma, obese asthmatic subjects have a relative abundance of Bacteroides (54%) and Firmicutes (26%). Notably, both phyla are part of the gastrointestinal microbiome, suggesting inoculation through gastroesophageal reflux which may be more common in obese individuals. Asthmatics identified as having improvement in their asthma control following treatment with inhaled corticosteroids appear to have a greater relative abundance of Actinobacteria (79.8%) in their airways relative to other asthmatics. Actinobacteria have been associated with the production of anti-inflammatory proteins and are speculated to be involved in increasing steroid responsiveness. Other studies have demonstrated that oral administration of probiotics, including Bifidobacterium species within the phyla Actinobacteria, lead to reduced Th2 cytokine production and eosinophilic inflammation, along with promotion of Regulatory T-cell (Treg) populations within the airway. We hypothesize that administration of over the counter oral probiotics containing Actinobacteria (Bifidobacterium) to obese asthmatic subjects will result in decreased airway inflammation and better asthma control by immune modulation.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe asthma requiring medium to high dose inhaled corticosteroids

   1. Patients will be recruited through the UAB Asthma Clinic and using the UAB Asthma Clinic Database for the Biospecimen Repository
   2. Patients must show spirometry with positive bronchodilator reversibility or have a positive Methacholine Challenge Test within 3 years of enrollment
2. Obesity as defined as BMI over 30
3. Self-reported or radiographic evidence of gastroesophageal reflux disease
4. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Inability of the subject to provide informed consent
2. Inability of the subject to undergo bronchoscopy
3. Use of monoclonal antibody within three months prior to enrollment
4. Use of immunosuppressive medication
5. Use of oral corticosteroids or antibiotics 4 weeks prior to enrollment
6. Use of anticoagulants (warfarin/Coumadin and heparin products).
7. Use of aspirin and/or other non-steroidal anti-inflammatory drugs or clopidogrel (Plavix) within 5 days of bronchoscopy.
8. Pregnancy
9. Diagnosis of HIV, active cancer, or liver disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
A change in the relative abundance of bifidobacterium species found in the airway. | 4 weeks
  The relative abundance of bacterial species in the airways of participants will be quantified from samples obtained during bronchoscopy and compared at baseline and after using oral probiotic supplements daily.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with researchers not included on the approved IRB

REFERENCES:
- [Background] Hilty M, Burke C, Pedro H, Cardenas P, Bush A, Bossley C, Davies J, Ervine A, Poulter L, Pachter L, Moffatt MF, Cookson WO. Disordered microbial communities in asthmatic airways. PLoS One. 2010 Jan 5;5(1):e8578. doi: 10.1371/journal.pone.0008578. PMID 20052417
- [Background] Huang YJ, Nariya S, Harris JM, Lynch SV, Choy DF, Arron JR, Boushey H. The airway microbiome in patients with severe asthma: Associations with disease features and severity. J Allergy Clin Immunol. 2015 Oct;136(4):874-84. doi: 10.1016/j.jaci.2015.05.044. Epub 2015 Jul 26. PMID 26220531
- [Background] Marri PR, Stern DA, Wright AL, Billheimer D, Martinez FD. Asthma-associated differences in microbial composition of induced sputum. J Allergy Clin Immunol. 2013 Feb;131(2):346-52.e1-3. doi: 10.1016/j.jaci.2012.11.013. Epub 2012 Dec 23. PMID 23265859
- [Background] Huang YJ, Nelson CE, Brodie EL, Desantis TZ, Baek MS, Liu J, Woyke T, Allgaier M, Bristow J, Wiener-Kronish JP, Sutherland ER, King TS, Icitovic N, Martin RJ, Calhoun WJ, Castro M, Denlinger LC, Dimango E, Kraft M, Peters SP, Wasserman SI, Wechsler ME, Boushey HA, Lynch SV; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. Airway microbiota and bronchial hyperresponsiveness in patients with suboptimally controlled asthma. J Allergy Clin Immunol. 2011 Feb;127(2):372-381.e1-3. doi: 10.1016/j.jaci.2010.10.048. Epub 2010 Dec 30. PMID 21194740
- [Background] Chang P, Friedenberg F. Obesity and GERD. Gastroenterol Clin North Am. 2014 Mar;43(1):161-73. doi: 10.1016/j.gtc.2013.11.009. Epub 2013 Dec 27. PMID 24503366
- [Background] MacSharry J, O'Mahony C, Shalaby KH, Sheil B, Karmouty-Quintana H, Shanahan F, Martin JG. Immunomodulatory effects of feeding with Bifidobacterium longum on allergen-induced lung inflammation in the mouse. Pulm Pharmacol Ther. 2012 Aug;25(4):325-34. doi: 10.1016/j.pupt.2012.05.011. Epub 2012 Jun 13. PMID 22705947